CLINICAL TRIAL: NCT04423874
Title: The Effect of Exposure to Aversive Non-verbal Vocalizations on Pain Tolerance
Acronym: CRYPAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Laboratoire ENES-CNPS (Université Lyon/Saint Etienne) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19CH215; 2020-A00274-35 (Other: ANSM)
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: nonverbal vocal communication; babies cries; pain tolerance; cold pressor test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy adult population aged 18 to 60 years. (Experimental): Their pain tolerance will be tested using the Cold Pressor Task while listening to vocalisations. Physiological measures will be taken using two techniques: Nociception Level Index and video pupillometry.
  Interventions: Behavioral: Cold pressor task (CPT); Diagnostic Test: index NOL; Behavioral: Playback Experiments; Diagnostic Test: Video-pupillometry

INTERVENTIONS:
Behavioral: Cold pressor task (CPT) — The cold pressor test is among the most common and established methods for studying human reactions to pain and pain tolerance.
  Participants submerge a hand in cold water (approx. 5°C) and are asked to keep their hand submerged for as long as can (until the sensation is intolerable), up to a maximum of 5 min.
  The procedure is safe because the hand is removed before adverse effects can occur.
  The participant will be given a break of 5 min in between trials, and will interchange hands between trials.
  During this break hand may to be place in warm water (25-35°C) for up to 4 min to normalise hand temperature, which will be measured before and after each trial using a digital thermometer held firmly in the palm of the hand. Each participant will complete no more than three trials (conditions) in a randomised order.
Diagnostic Test: index NOL — Measurement of the index NOL™: Four sensors, placed non-invasively on one of the four participants' fingers, will make it possible to calculate a dozen physiological parameters converts in real time into a pain index called NOL (for Nociception Level Index).
Behavioral: Playback Experiments — During the experience, participants are led to listen, via headphones, to aversive non-verbal vocalizations (baby crying). The sound levels used to broadcast the non-verbal vocalisations will be scrupulously measured using approved and certified equipment during the preparation of the experiments. These sound volumes will be chosen so as not to inconvenience participants.
Diagnostic Test: Video-pupillometry — This technique is based on the observation of the dilatation of the pupil during the perception of a nociceptive stimulus in test persons.

SUMMARY:
Humans produce non-verbal vocalizations (shouting, growling, screaming), laughter, ...) in various contexts that are likely to perform biological functions.

and important social issues. Yet despite their importance in the human vocal repertoire, the mechanisms and functions of non-verbal vocalizations remain little studied and poorly understood including in humans.

In this context, the investigators wish to examine how the perception of vocalizations non-verbal aversive behaviours influence pain tolerance in healthy adults.

DETAILED DESCRIPTION:
Humans produce nonverbal vocalisations such as screams, grunts, roars, cries and laughter across a variety of contexts. Yet despite the prominence and apparent importance of these nonverbal sounds in human communication, the investigators still know very little about their influence on human perception and behaviour. That's why, in this study, the investigators will examine specifically the influence of nonverbal vocal perception on pain tolerance.

The remainder of the study will involve up to three trials of a pain tolerance (cold pressor) task, during which the investigators will ask participants to listen to vocalisations (e.g., babies' cries or babbling) while submerging the participant's hand in bath of circulating cold water.

The results of the study will contribute to theoretical understanding of the functions of nonverbal vocal communication in humans, in particular the influence of nonverbal vocal and perception (of babies' cries) on pain tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Participant in good health
* Affiliated or entitled participant in a social security scheme
* Participant who received informed information about the study and co-signed, with the investigator, a consent to participate in the study

Exclusion Criteria:

* Chronic pain
* High blood pressure or poor circulation
* Cardiac or vascular disease, or a heart condition (including symptoms of Raynaud's syndrome)
* Allergy or hypersensitivity to cold
* Diabetes
* Epilepsy
* Pregnancy
* Recent serious injury
* Neurological or psychiatric condition known to affect pain tolerance (e.g., peripheral neuropathy, schizophrenia)
* History of fainting or seizures
* History of frostbite

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Pain tolerance | at inclusion
  Delay (in seconds) in removing the hand when testing the Cold Pressor.

SECONDARY OUTCOMES:
Onset of pain | at inclusion
  Participant verbally indicates when he or she begins to feel the sensation of pain (time of onset measured in seconds).
Pain intensity | at inclusion
  Subjective assessment of maximum pain intensity by participants for a given trial.
  Measured by scale of 0 (no pain) at 100 (extreme pain).
Correlation between NOL index and video pupillometry results | at inclusion
  Measurement of the NOL index (index ranging from 0 to 100) and measurement of pupillary diameter and its variations (in mm) in response to nociceptive stimuli by video pupillometry.

CONTACTS AND LOCATIONS:
Overall Officials: Roland PEYRON, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Centre Hospitalier Universitaire SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No